CLINICAL TRIAL: NCT00005481
Title: Epidemiology of Impaired Coagulant Balance in Diabetes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4965; R01HL058329 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus; Blood Coagulation Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus; Blood Coagulation Disorders

SUMMARY:
To determine the nature, extent and molecular mechanisms responsible for impaired fibrinolysis in White, Black, Hispanic and American Indian populations with respect to the presence or absence of diabetes. The overall objective is to determine whether impairments of fibrinolysis underlie subclinical and clinical vascular disease in diabetes in specific populations with and without accelerated microvascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

The results of this project should clarify the extent to which results obtained in experimental animals pertain directly to diabetes in human subjects. The study will also assist in the interpretation of results from clinical studies and from platelet activation experiments.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Tracy — University of Vermont

REFERENCES:
- [Background] Tracy RP. Inflammation markers and coronary heart disease. Curr Opin Lipidol. 1999 Oct;10(5):435-41. doi: 10.1097/00041433-199910000-00008. PMID 10554706
- [Background] Smiles AM, Macy EM, Sakkinen PA, Bovill EG, Mann KG, Tracy RP. Variability in plasma prothrombin concentration: implications for use in epidemiology. Blood Coagul Fibrinolysis. 1998 Sep;9(6):525-31. doi: 10.1097/00001721-199809000-00010. PMID 9819003
- [Background] Festa A, D'Agostino R Jr, Tracy RP, Haffner SM; Insulin Resistance Atherosclerosis Study. Elevated levels of acute-phase proteins and plasminogen activator inhibitor-1 predict the development of type 2 diabetes: the insulin resistance atherosclerosis study. Diabetes. 2002 Apr;51(4):1131-7. doi: 10.2337/diabetes.51.4.1131. PMID 11916936
- [Background] Lewis MR, Callas PW, Jenny NS, Tracy RP. Longitudinal stability of coagulation, fibrinolysis, and inflammation factors in stored plasma samples. Thromb Haemost. 2001 Dec;86(6):1495-500. PMID 11776319
- [Background] Festa A, D'Agostino R Jr, Williams K, Karter AJ, Mayer-Davis EJ, Tracy RP, Haffner SM. The relation of body fat mass and distribution to markers of chronic inflammation. Int J Obes Relat Metab Disord. 2001 Oct;25(10):1407-15. doi: 10.1038/sj.ijo.0801792. PMID 11673759
- [Background] Hanley AJ, Karter AJ, Festa A, D'Agostino R Jr, Wagenknecht LE, Savage P, Tracy RP, Saad MF, Haffner S; Insulin Resistance Atherosclerosis Study. Factor analysis of metabolic syndrome using directly measured insulin sensitivity: The Insulin Resistance Atherosclerosis Study. Diabetes. 2002 Aug;51(8):2642-7. doi: 10.2337/diabetes.51.8.2642. PMID 12145182
- [Background] Festa A, D'Agostino R Jr, Tracy RP, Haffner SM. C-reactive protein is more strongly related to post-glucose load glucose than to fasting glucose in non-diabetic subjects; the Insulin Resistance Atherosclerosis Study. Diabet Med. 2002 Nov;19(11):939-43. doi: 10.1046/j.1464-5491.2002.00824.x. PMID 12421431
- [Background] Festa A, D'Agostino R Jr, Rich SS, Jenny NS, Tracy RP, Haffner SM. Promoter (4G/5G) plasminogen activator inhibitor-1 genotype and plasminogen activator inhibitor-1 levels in blacks, Hispanics, and non-Hispanic whites: the Insulin Resistance Atherosclerosis Study. Circulation. 2003 May 20;107(19):2422-7. doi: 10.1161/01.CIR.0000066908.82782.3A. Epub 2003 Apr 28. PMID 12719278